CLINICAL TRIAL: NCT03332147
Title: Clinical Evaluation of the RHEA Vital Sign Vigilance System in Hospital Patients
Brief Title: Clinical Evaluation of the RHEA Vital Sign Vigilance System in Hospital Patients Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Darma Inc. (Industry)
Collaborators: Tufts Medical Center (Other); Medstar Health Research Institute (Other); Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Screening
Other Study IDs: RHEA EL30-2017-001
Record Dates: First submitted 2017-10-27; First posted 2017-11-06 (Actual); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Vital Sign Monitoring

STUDY DESIGN:
Intervention Model Description: The reference device and Patient Monitor are used to monitor the heart rate (HR) and respiratory rate (RR) of the same participant at the same time in Test 1. The RHEA device and patient monitor are used to monitor the heart rate and respiratory rate of the same participant at the same time in Test 2. The two tests results will be compared and evaluated for the accuracy of the two devices. The RHEA device is used alone to evaluate the accuracy of motion or no motion alarm in Test 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Investigational Group (Experimental): The RHEA device and Patient Monitor Device are used to monitor the heart rate (HR) and respiratory rate (RR) of participants.
  Interventions: Device: Investigational Group
- reference group-Earlysense system (Active Comparator): The reference device and Patient Monitor Device are used to monitor the heart rate (HR) and respiratory rate (RR) of participants.
  Interventions: Device: reference group-Earlysense system

INTERVENTIONS:
Device: Investigational Group — The RHEA device and Philips Patient Monitor MX400 are used to monitor the heart rate (HR) and respiratory rate (RR) of participants.
  Arms: Investigational Group
Device: reference group-Earlysense system — The reference device Earlysense 2.0 system(vital sign monitoring system) and Philips Patient Monitor MX400 are used to monitor the heart rate (HR) and respiratory rate (RR) of participants.
  Arms: reference group-Earlysense system

SUMMARY:
This study compares both of the investigational device and reference device to the gold standard Patient Monitor of the accuracy of heart rate and respiratory rate monitoring. The primary variables for the analysis of heart rate (HR) and respiratory rate (RR) are each of the overall mean roots mean square difference (RMSD). Results of the investigational device and reference device compared with the patient monitor is evaluated to see if there are equivalent. Motion and bed exit accuracy will be evaluated by comparing with the manual observation.

DETAILED DESCRIPTION:
The testing will be conducted in three periods. In the Accuracy Tests (periods

1 and 2), one of the contact-free devices will be used to monitor the HR and RR, while being compared with the Patient Monitor. The RHEA investigational device and reference device will be used to monitor the same subject at different times, as the sensors of the two devices are placed at a similar location of the bed. HR and RR will be recorded for all three devices.

The primary hypotheses for HR, are as follows:

Adults HO: μ = 3.25 vs. HA: μ < 3.25

The primary hypotheses for RR, are as follows:

Adults HO: μ = 2.25 vs. HA: μ < 2.25 where μ represents the population mean HR or RR. If the upper bound of the confidence interval is less than the hypothesized value, the corresponding null hypothesis will be rejected. Comparison of the performance of the two contract-free devices will be performed on the recorded results via statistical analysis. The hypothesis here is that the two devices have equivalent performance. The third test will assess the ability of the RHEA device to accurately detect motion in or exit from the bed, as compared to the manual observation. Motion and no motion accuracy will each be calculated along with their respective two-sided 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 years old and above.
2. Provide written informed consent.
3. Weight ranging from 20 to 150 kg inclusive.
4. Are located in a non-ICU hospital setting.
5. Agree to not eat during the testing period.
6. Agree to keep still.

Exclusion Criteria:

1. Are connected to a device which may interfere with the device monitoring in this study.
2. Are receiving any bedside care which may be incompatible with the study procedures.
3. Sleep apnea.
4. Pregnant or breastfeeding.
5. A likely need to receive or undergo a procedure during the testing period.
6. Cannot accept a nasal cannula, or have a monitor lead placed on the chest.
7. A significant medical condition in the judgement of the investigator, which may compromise the study testing procedures.
8. Are wearing pacemaker or defibrillator.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2017-11-04 (Actual); Primary Completion 2018-05-25 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
RMSD of Investigational Device's Heart Rate and Gold Standard Device's heart rate | 45 days
  Record 20 valid pair heart rate displayed in the investigational device and patient monitor at the same time every one minutes.Calculate the root mean square difference(RMSD) of the heart rate for the investigational device and the gold standard device.
RMSD of Investigational Device's Respiratory Rate and Gold Standard Device's Respiratory rate | 45 days
  Record 20 valid pair respiratory rate displayed in the investigational device and patient monitor at the same time every one minutes.Calculate the root mean square difference(RMSD) of the respiratory rate for the investigational device and the gold standard device.

SECONDARY OUTCOMES:
Heart Rate t Test Comparison result between the Investigational Device and the Reference Device | 45 days
  Record 20 valid heart rate displayed in the reference device and patient monitor at the same time every one minute.
  Calculate the t test results for heart rate for the reference device and the investigational device.
Respiratory Rate t Test Comparison result between the Investigational Device and the reference device | 45 days
  Record 20 valid respiratory rate displayed in the reference device and patient monitor at the same time every one minute. Calculate the t test results for respiratory rate for the reference device and the investigational device.
Motion Notification Accuracy(%) | 45 days
  Record the time for each instructed movements from manual observation and time for movements notification shown in the investigational device. Calculate the times matched between these two to get the accuracy.
Bed Exit Notification Accuracy(%) | 45 days
  Record the time for each instructed bed exit from manual observation and time for bed exit notification shown in the investigational device. Calculate the times matched between these two to get the accuracy.

CONTACTS AND LOCATIONS:
Overall Officials: Judith Cullinane, MSN, Principal Investigator — Tufts Medical Center; Arrel Olano, MD, Principal Investigator — Medstar Health Research Institute; Rehan Qayyum, MD, Principal Investigator — Virginia Commonwealth University
Locations (3):
- United States (3):
  - Medstar Health Research Institute, Washington D.C., District of Columbia
  - Tufts Medical Center, Boston, Massachusetts
  - Virginia Commonwealth University, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-23): https://cdn.clinicaltrials.gov/large-docs/47/NCT03332147/Prot_SAP_000.pdf